CLINICAL TRIAL: NCT02894099
Title: Blood Glucose, Insulin Response and Inflammatory Markers in Sedentary Elderly During Prolonged Sitting Time Versus Intermittent Sitting Time
Brief Title: Cardiovascular Risk in Sedentary Elderly During Prolonged Sitting Time Versus Intermittent Sitting Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Ferriolli, Assistant professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1563/2015
Record Dates: First submitted 2016-07-26; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Sedentary Lifestyle
Keywords: Aged; Sedentary Behaviour; Blood Glucose; Insulin; Inflammatory markers
MeSH Terms: conditions — Sedentary Behavior; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prolonged Sitting Time (PST) (Experimental): Uninterrupted sitting time of 5 hours
  Interventions: Other: Prolonged sitting time
- PST+Light intensity Short bouts PA (Experimental): Sitting prolonged interrupted with breaks of 2 minutes of light physical activity
  Interventions: Other: PST+Light intensity Short bouts PA
- PST+Moderate intensity Short bouts PA (Experimental): Sitting prolonged interrupted with breaks of 2 minutes of moderate physical activity
  Interventions: Other: PST+Moderate intensity Short bouts PA
- PST+Moderate intensity Long bouts PA (Experimental): Sitting prolonged interrupted with breaks of 10 minutes of moderate physical activity
  Interventions: Other: PST+Moderate intensity Long bouts PA

INTERVENTIONS:
Other: Prolonged sitting time — Volunteers will be continuously sitting on a chair for 5 hours and should move the least possible. If the participant needs to stand from the chair, the stage will be invalidated.
  Arms: Prolonged Sitting Time (PST)
Other: PST+Light intensity Short bouts PA — Volunteers will have their time sitting interrupted every 20 minutes for 2 minutes of physical activity of low intensity. In the active period, participants will be encouraged to walk in the hallway and reach a training heart rate between 50-60% HR max predicted for the age and measured by heart rate monitor. The Borg scale will be used at the beginning and the end of each active period in order to measure the subjective effort of the participants. In the end the volunteers will be sitting 5 hours and have 30 minutes (15 bouts of 2 minutes) of light intensity physical activity.
  Arms: PST+Light intensity Short bouts PA
Other: PST+Moderate intensity Short bouts PA — Volunteers will have their time sitting interrupted every 20 minutes for 2 minutes of physical activity of moderate intensity. In the active period, participants will be encouraged to walk in the hallway and reach a training heart rate between 65 a 75% HR max predicted for the age and measured by heart rate monitor. The Borg scale will be used at the beginning and the end of each active period in order to measure the subjective effort of the participants. In the end the volunteers will be sitting 5 hours and have 30 minutes (15 bouts of 2 minutes)of moderate intensity physical activity.
  Arms: PST+Moderate intensity Short bouts PA
Other: PST+Moderate intensity Long bouts PA — Volunteers will have their time sitting interrupted every 75 minutes for 10 minutes of physical activity of moderate intensity. In the active period, participants will be encouraged to walk in the hallway and reach a training heart rate between 65 a 75% HR max predicted for the age and measured by heart rate monitor. The Borg scale will be used at the beginning and the end of each active period in order to measure the subjective effort of the participants. In the end the volunteers will be sitting 5 hours and have 30 minutes (3 bouts of 10 minutes) of moderate intensity physical activity.
  Arms: PST+Moderate intensity Long bouts PA

SUMMARY:
In adults, the sedentary behavior was related to cardiovascular risk markers, regardless of the level of physical activity (PA). However, the interruption of prolonged sedentary time has shown positive results even when performed in breaks of low intensity and short duration of activity. The aim of this study is to analyze the influence of a sedentary uninterrupted period, as well as different forms of breaks in sedentary time for the glycemic, insulin and inflammatory markers responses in older adults. This is a controlled clinical trial to be conducted in older (≥ 65 years) and sedentary (<150 min / week of moderate to vigorous physical activity) people. Those with BMI ≥ to 35.00 kg /m2; diabetic, on medication for glycemic control, or with absolute or relative contraindications to PA practice will not be included . Participants will undergo four phases of intervention separated by an interval of 7 days: (1) Prolonged Sitting Time(PST), in which older people will stay for 5 hours seated; (2) Prolonged sitting with PA of light intensity and short duration (LiSd), time sitting is interrupted for PA bouts of 50-60% of the Heart Rate (HR)max; (3) Prolonged sitting with PA of moderate intensity and short duration (MiSd), time sitting will be interrupted for PA bouts of 65-75% predicted HR max; (4) Prolonged sitting with PA of moderate intensity and long duration (MiLd,) time sitting will be interrupted with PA bouts of 65-75% of HRmax. PA bouts will be performed by walking into a hallway every 20 minutes of sitting time and will last 2 minutes, except in MiLd phase (10 minute breaks every 75 minutes). To evaluate the effects of different PA interruptions in plasma glucose, serum insulin and inflammatory markers, blood samples will be collected serially (-30min, Baseline and 30min, 1h, 2h, 3h, 4h and 5h after a standardized meal. It is expect that interruption of sedentary time, even with breaks of short duration and light intensity can bring benefits to cardiovascular risk markers even in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary older women according World Health Organization, defined as not performing moderate to vigorous physical activity and vigorous for 150 min / week for at least 3 months;
* BMI <to 35.00 kg / m2;
* Sign the Informed Consent.

Exclusion Criteria:

* Previous diagnosis of Diabetes Mellitus;
* Use of any medication for glycemic control;
* Orthopedic problems that impair walking or use of orthoses for walking.
* Relative or absolute contraindications to perform physical activity.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose area under curve during 5 hours in four different phases of intervention | 4 weeks
  Assessed by serial blood sampling.The first blood sampling is performed 30 minutes before ingestion of a standard meal mixed solution composed of carbohydrate, fat and protein. The collection of serial blood will be collected in time (-30min, Baseline, 30min, 1h, 2h, 3h, 4h and 5h after the meal). The results will be expressed in mg.dl.
Change in insulin area under curve during 5 hours in four different phases of intervention | 4 weeks
  Assessed by serial blood sampling. The first blood sampling is performed 30 minutes before ingestion of a standard meal mixed solution composed of carbohydrate, fat and protein. The collection of serial blood will be collected in time (-30min, Baseline, 30min, 1h, 2h, 3h, 4h and 5h after the meal).The results will be expressed in µIU/ml.

SECONDARY OUTCOMES:
Assessment of physical performance | 1 day
  The physical performance will be evaluated by the Short Physical Performance Battery test.
Assessment of handgrip strength | 1 day
  Measure of handgrip strength with a manual dynamometer (Saehan)
Assessment of muscle strength of knee extensors | 1 day
  Measure of muscle strength of the lower limbs (knee extension) with a isokinetic dynamometer (Biodex 4 Pro)
Physical Activity behaviour | 7 days
  use of a tri-axial accelerometer to measure profile of spontaneous physical activity
Change in Inflammatory Cytokines area under curve during 5 hours in four different phases of intervention | 4 weeks
  Assessed by serial blood sampling. The first sampling is performed 30 minutes before ingestion of a standard meal mixed solution composed of carbohydrate, fat and protein. The collection of serial blood will be collected in time (-30min, Baseline, 30min, 1h, 2h, 3h, 4h and 5h after the meal).

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ferriolli, PhD, Principal Investigator — USao Paulo
Locations (1):
- Clinics Hospital of the Ribeirao Preto Medical School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- [Background] Benatti FB, Ried-Larsen M. The Effects of Breaking up Prolonged Sitting Time: A Review of Experimental Studies. Med Sci Sports Exerc. 2015 Oct;47(10):2053-61. doi: 10.1249/MSS.0000000000000654. PMID 26378942
- [Background] Bailey DP, Locke CD. Breaking up prolonged sitting with light-intensity walking improves postprandial glycemia, but breaking up sitting with standing does not. J Sci Med Sport. 2015 May;18(3):294-8. doi: 10.1016/j.jsams.2014.03.008. Epub 2014 Mar 20. PMID 24704421
- [Background] Chastin SF, Egerton T, Leask C, Stamatakis E. Meta-analysis of the relationship between breaks in sedentary behavior and cardiometabolic health. Obesity (Silver Spring). 2015 Sep;23(9):1800-10. doi: 10.1002/oby.21180. PMID 26308477
- [Background] Bailey DP, Broom DR, Chrismas BC, Taylor L, Flynn E, Hough J. Breaking up prolonged sitting time with walking does not affect appetite or gut hormone concentrations but does induce an energy deficit and suppresses postprandial glycaemia in sedentary adults. Appl Physiol Nutr Metab. 2016 Mar;41(3):324-31. doi: 10.1139/apnm-2015-0462. Epub 2015 Dec 14. PMID 26872294
- [Background] Dunstan DW, Wiesner G, Eakin EG, Neuhaus M, Owen N, LaMontagne AD, Moodie M, Winkler EA, Fjeldsoe BS, Lawler S, Healy GN. Reducing office workers' sitting time: rationale and study design for the Stand Up Victoria cluster randomized trial. BMC Public Health. 2013 Nov 9;13:1057. doi: 10.1186/1471-2458-13-1057. PMID 24209423